CLINICAL TRIAL: NCT06597058
Title: A Double-Blind, Placebo-Controlled Phase 2 Estimation Study of Fixed Dose Drugs Combination Type of Polypill Administered to Subjects With Alzheimer's Disease
Brief Title: Phase 2 Estimation Study of Fixed Dose Drugs Combination Type of Polypill
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Noah Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T000439
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Neurodegeneration; Cognitive Impairments; Mental Deterioration; Loss of Memory
MeSH Terms: conditions — Alzheimer Disease; Dementia; Nerve Degeneration; Cognitive Dysfunction; Amnesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAR COMBO (Experimental): MAR Active 0.6 g, Tablet, once-daily, 180 days
  Interventions: Drug: MAR
- MAR PLACEBO (Placebo Comparator): MAR Placebo 0.6 g, Tablet, once-daily, 180 days
  Interventions: Drug: MAR

INTERVENTIONS:
Drug: MAR — Once-daily tablet

SUMMARY:
This is an estimation-focused Phase 2 study designed to explore and quantify treatment-related changes across multiple clinical outcomes in patients with Alzheimer's disease over a 210-day period. The anticipated study population are males and females aged 50-85 years with very mild to severe Alzheimer's Disease. The duration of individual patient participation will be approximately 224 Days: up to 14 days for Screening, 180 days for study drug administration, and a final follow-up visit at 210 days. The planned study duration is 12-18 months from Screening of the first patient until the last follow-up of the last patients.

ELIGIBILITY:
Inclusion Criteria:

1. Prior diagnosis of mild-to-severe cognitive impairment or probable AD according to the National Institute on Aging and the Alzheimer's Association guidelines by a qualified health practitioner;
2. History of cognitive and functional decline over at least 1 year that is either documented in medical records or by history from an informant who knows the patient well;
3. Male or female, age 50 to 85 years (inclusive) at the Screening Visit;
4. Patient must be ambulatory and reside with a reliable, competent adult (study partner) who may or may not also be the patient's legally authorized representative (LAR) for informed consent;
5. Patient must be able to swallow the study medication (without any alteration to the tablet like crushing, cutting in half, or dissolving in a liquid);
6. Body weight at screening is ≥40kg;
7. CDR-SB of 3.0 or higher at Screening Visit;
8. MMSE-2 ≥8 and≤24 at the Screening Visit;
9. Patient must be able to understand the nature of the study and have the opportunity to have any questions answered and provide their consent. In the absence of patient's ability to provide informed consent, the informed consent must be obtained from the patient's Legally Authorized Representative (LAR);
10. For patients receiving an anticholinesterase inhibitor, memantine, or herbal medication for AD, the dose must have been stable for at least 3 months prior to the Screening Visit, and patient must agree to maintain this dose for the duration of the study;
11. Patients currently treated with a statin must agree to stop their statin therapy for the duration of treatment (180 days);
12. Creatinine Clearance >30 mL/min at Screening;
13. Negative HIV and HCV test at Screening;
14. Complete blood count (CBC), blood chemistry, serum cholesterol, triglycerides, thyroid-stimulating hormone (TSH), and urinalysis, within normal reference ranges or not clinically significant as assessed by the Investigator at Screening;
15. Physical examination, vital signs, and ECG within normal ranges or not clinically significant as assessed by the Investigator at Screening;
16. Female patients may participate if they meet 1 of the following criteria:

    1. Surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or
    2. Post-menopausal, defined as
    3. Permanent cessation of menstruation for ≥12 months without an alternative medical cause (regardless of follicle-stimulating hormone [FSH] value) at the Screening Visit, or
    4. Cessation of menstruation for <12 months and FSH >40 mIU/mL at the Screening Visit.

    Note: Patients with persistent menses due to hormonal therapy may participate if a urine pregnancy test (UPT) at the Screening Visit is negative and they agree to continued testing at every study visit.
17. Male patients must agree to use a barrier method of contraception and refrain from donating sperm for the duration of their participation in the study and for 2 months thereafter.

Exclusion Criteria:

1. Patient has had a myocardial infarction, unstable angina, stroke, transient ischemic attack or required intervention for any of these conditions (e.g., coronary artery bypass graft, percutaneous coronary intervention via cardiac catheterization, thrombolytic therapy) within 6 months of the Screening Visit;
2. Has other neurological disorders, including vascular dementia, Parkinson's disease, frontotemporal dementia, Huntington's disease, amyotrophic lateral sclerosis, multiple sclerosis, progressive supranuclear palsy, neurosyphilis, dementia with Lewy bodies, other types of dementia, mental retardation, hypoxic cerebral damage, and cognitive impairment from head trauma;
3. Scheduled or anticipates vaccination with a live vaccine during the study;
4. Current use of a cannabidiol or derivative;
5. Current use of digoxin;
6. Acute or chronic liver disease;
7. AST >1.5 times the Upper Limit of Normal
8. ALT > 1.5 times the Upper Limit of Normal
9. Schizophrenia, bipolar disorder, suicidal ideation, major depression, or delirium; Note: Stable (>2 years) treated depression without suicidal ideation is acceptable;
10. Current therapy with a tetracycline;
11. Current therapy with sirolimus or a rapalog macrolide antibiotic;
12. Known allergies to any of the active drugs: tetracycline antibiotics, rapalog macrolide antibiotics, or statin therapies;
13. Treatment with another investigational drug, device, or intervention within 30 days prior to the Screening Visit;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Dementia Rating - Global Score | Day 210
  CDR - Global Score: To estimate the magnitude and variability of clinical response to a drug combination Tablet in patients with Alzheimer's disease (AD) after 180 days of treatment against Placebo Tablet.
  The CDR scale is a widely used dementia staging instrument that produces a global score. This study will use global score for estimation, comparisons and analysis. The global score ranges from 0 to 3. The sites are instructed to use a standardized online calculator for scoring. This resulting calculation reflects the following scoring 0 = normal, no cognitive impairment; 0.5 = very mild dementia, minimal impairment in one domain; 1 = mild dementia, noticeable impairment in one or more domains; 2 = moderate dementia, significant impairment in multiple domains; 3 = severe dementia, major impairment in multiple domains.
Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score | Day 210
  CDR - SB: To estimate the magnitude and variability of clinical response to a drug combination Tablet in patients with Alzheimer's disease (AD) after 180 days of treatment against Placebo Tablet. The CDR scale is a widely used dementia staging instrument that produces a summated score (sum of boxes score). This study will use the summated score, comparisons and analysis. The "Sum of boxes" scoring methodology sums the score for each of the 6 domains and provides a value ranging from 0 to 18 that can change in of 0.5 or greater. Higher scores indicate greater disease severity. A positive change from baseline indicates clinical decline. Score Range from 0 to 18. Response choices are 0 = normal; 0.5 to 2.5 = questionable impairment; 3.0 to 4.0 = very mild dementia; 4.5 to 9.0 = mild dementia; 9.5 to 15.5 = moderate dementia; 16.0 to 18.0 = severe dementia.
Mini-Mental Scale Evaluation, 2nd Edition (MMSE-2) Score | Day 210
  MMSE-2: To estimate the magnitude and variability of clinical response to a drug combination Tablet in patients with Alzheimer's disease (AD) after 180 days of treatment against Placebo Tablet. The MMSE-2 is a widely used test of cognitive function among the elderly. The Standard Version consists of a 30-point questionnaire that includes tests of orientation, attention, memory, language, and visual-spatial skills. Score Range from 0 to 30. Response choices are 30 = normal; 26 to 29 = mild cognitive impairment; 21 to 25 = early stage dementia or mild cognitive impairment; 11 to 20 = middle stage dementia or moderate cognitive impairment; 0 to 10 = late stage dementia or severe cognitive impairment.
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-COG) | Day 210
  ADAS-COG: To estimate the magnitude and variability of clinical response to a drug combination Tablet in patients with Alzheimer's disease (AD) after 180 days of treatment against Placebo Tablet. The ADAS-COG is used to assess cognitive symptoms of dementia. It consists of 7 performance items and 4 clinician-rated items assessing memory, orientation, language and praxis. Score Range from 0 to 70. Response choices are 0 to 10 = minimal to no cognitive impairment; 11 to 20 = mild cognitive impairment; 21 to 30 = moderate cognitive impairment; 31 to 70 = severe cognitive impairment.
Alzheimer's Disease Cooperative Study-ADL scale (ADCS-ADL) | Day 210
  ADCS-ADL: To estimate the magnitude and variability of clinical response to a drug combination Tablet in patients with Alzheimer's disease (AD) after 180 days of treatment against Placebo Tablet. The ADCS-ADL is a comprehensive battery of ADL questions used to measure the functional capabilities of patients; each item is rated from the highest level of independent performance to complete loss. Score Range from 0 to 78. Response choices are 0 to 20 = severe impairment; 21 to 40 = moderate impairment; 41 to 60 = mild impairment; 61 to 78 = minimal impairment.
Clinical Global Impressions - Improvement (CGI-I) | Day 210
  CGI-I: To estimate the magnitude and variability of clinical response to a drug combination Tablet in patients with Alzheimer's disease (AD) after 180 days of treatment against Placebo Tablet. The Clinical Global Impressions-Improvement (CGI-I) scale will be assessed at all visits after Baseline. The Investigator (or designee) will answer the following question: "Compared to the patient's condition at Baseline. Score Range from 1 to 7. Response choices are: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change from Baseline; 5 = minimally worse; 6 = much worse; 7 = very much worse since Baseline".
Clinical Global Impressions - Severity (CGI-S) | Day 210
  CGI-S: To estimate the magnitude and variability of clinical response to a drug combination Tablet in patients with Alzheimer's disease (AD) after 180 days of treatment against Placebo Tablet. The Clinical Global Impressions-Severity (CGI-S) scale will be assessed at Baseline and all visits afterward. The Investigator (or designee) will answer the following question: "Considering your total clinical experience with AD, how ill is the patient at this time?" Score Range from 1 to 7. Response choices are 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients.
Clinical Dementia Rating - Global Score (Exploratory) | Day 210
  Change from Baseline in the Clinical Dementia Rating - Global Score after 210 days (Global Score ranges from 0 to 3; a lower score indicates no disease; a higher score indicates greater disease severity; 0 = normal, 3 = severe dementia)
Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score (Exploratory) | Day 210
  Change from Baseline in CDR-SB Score after 210 days (CDR-SB Score ranges from 0 to 18; a lower score indicates no disease; a higher score indicates greater disease severity; 0 = normal, 18 = severe dementia)
Mini-Mental Scale Evaluation, 2nd Edition (MMSE-2) Score (Exploratory) | Day 210
  Change from Baseline from MMSE-2 Score through 210 days (MMSE-2 Score ranges from 0 to 30; a lower score indicates severe dementia; a higher score indicates better cognitive function; 0 to 10 = late stage dementia or severe cognitive impairment, 30 = normal)
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-COG) (Exploratory) | Day 210
  Change from Baseline in ADAS-COG Score through 210 days (ADAS-COG Score ranges from 0 to 70; a lower score indicates better cognitive function; a higher score indicates greater dysfunction; 0 to 10 = minimal to no cognitive impairment, 31 to 70 = severe cognitive impairment)
Alzheimer's Disease Cooperative Study-ADL scale (ADCS-ADL) (Exploratory) | Day 210
  Change from Baseline in ADCS-ADL Score through 210 days (ADCS-ADL Score ranges from 0 to 78; a lower score indicates greater severity; a higher score indicates better functioning in daily activities; 0 to 20 = severe impairment, 61 to 78 = minimal impairment)
Clinical Global Impressions - Improvement (CGI-I) (Exploratory) | Day 210
  Change from Baseline in CGI-I Score through 210 days (CGI-I Score ranges from 1 to 7; a lower score indicates the patient has improved; a higher score indicates the patient is very much worse since Baseline; 1 = very much improved, 7 = very much worse since Baseline)
Clinical Global Impressions - Severity (CGI-S) (Exploratory) | Day 210
  Change from Baseline in CGI-S Score through 210 days (CGI-S Score ranges from 1 to 7; a lower score indicates the patient is less severely ill; a higher score indicates among the most extremely ill patients; 1 = normal, not at all ill, 7 = among the most extremely ill patients)
Treatment-emergent adverse events (TEAEs) | Day 210
  Incidence of TEAEs through Day 210
Serious Adverse Events (SAEs) | Day 210
  Incidence of SAEs from informed consent through Day 210
Adverse Events (AEs) | Day 210
  Incidence of AEs from informed consent through Day 210

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Scottsdale Clinical Trials (Noah Clinical Site 017), Scottsdale, Arizona
  - Marvel Clinical Research (Noah Clinical Site 010), Huntington Beach, California
  - Accel Research Sites (Noah Clinical Site 019), DeLand, Florida
  - Health Awareness (Noah Clinical Site 020), Jupiter, Florida
  - Life Well Research Center (Noah Clinical Site 008), Miami, Florida
  - Regenerate Primary Medical Research (Noah Clinical Site 003), Miami, Florida
  - Miami Jewish Health (Noah Clinical Site 023), Miami, Florida
  - Neurology Associates of Ormond Beach (Noah Clinical Site 015), Ormond Beach, Florida
  - International Medical Investigational Centers (Noah Clinical Site 001), Palmetto Bay, Florida
  - Best Choice Medical and Research Service (Noah Clinical Site 025), Pembroke Pines, Florida
  - Denali Health Plant City, LLC (Noah Clinical Site 024), Plant City, Florida
  - Boston Clinical Trials (Noah Clinical Site 006), Boston, Massachusetts
  - IMA Clinical Research (Noah Clinical Site 004), Albuquerque, New Mexico
  - Carolina Research Center, Inc. (Noah Clinical Site 009), Shelby, North Carolina
  - Tekton Research (Noah Clinical Site 002), Yukon, Oklahoma
  - Olympus Clinical Research (Noah Clinical Site 014), Katy, Texas

IPD SHARING:
Plan to Share IPD: No